CLINICAL TRIAL: NCT06382337
Title: Maxillary Anterior Teeth Replacement With Immediate Dental Implants Utilizing Vestibular Socket Therapy Versus Ice Cream Cone Technique
Brief Title: Immediate Dental Implants in The Upper Anterior Region
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A03010240S
Record Dates: First submitted 2024-04-10; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Teeth Loss; Alveolar Bone Resorption
Keywords: VST; immediate dental implants; ice cream cone technique; Type 2 socket
MeSH Terms: conditions — Anodontia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A :immediate dental Implants cases with ice-cream cone technique in type 2 socket (Experimental): immediately placed implants in which the socket defect will be treated utilizing ice cream cone technique by Dennis Tarnow using collagen membrane , allograft bone graft and custom healing abutments
  Interventions: Other: Group A : ice cream cone technique
- Group B : immediate dental Implants cases with the vestibular socket therapy in type 2 socket (Experimental): 8 immediately placed implants in which the socket defect will be treated utilizing vestibular socket therapy technique using cortical lamina , allograft , bone tacks for fixation and custom healing abutment
  Interventions: Other: Group B : the vestibular socket therapy

INTERVENTIONS:
Other: Group A : ice cream cone technique — collagen membrane and allograft bone for labial plate augmentation simultaneously with immediate implants placements in maxillary anterior region in the defected type 2 socket , custom healing abutment for soft tissue preservation in ice cream cone group
  Arms: Group A :immediate dental Implants cases with ice-cream cone technique in type 2 socket
Other: Group B : the vestibular socket therapy — cortical lamina fixed by bone tacks and allograft bone for labial plate augmentation simultaneously with immediate implants placements in maxillary anterior region in the defected type 2 socket , custom healing abutment for soft tissue preservation in ice cream cone group
  Arms: Group B : immediate dental Implants cases with the vestibular socket therapy in type 2 socket

SUMMARY:
The aim of the study will be to evaluate maxillary anterior teeth replacement with immediate dental implant utilizing vestibular socket therapy versus ice cream cone technique both clinically and radiographically.

DETAILED DESCRIPTION:
Tooth loss is the endpoint of oral diseases, such as dental caries and periodontitis, and reflects the utilization of dental services during a lifetime .

The incidence of tooth loss has significantly declined at the global levels. However, tooth loss and oral diseases are still a major public health concern worldwide.

In the anterior region, the common reason for tooth loss is due to traumatic injury or congenital anomaly, loss of a single tooth may cause functional and esthetic deficits to the patient. Tooth extraction usually accompanies alveolar ridge resorption along with loss of preexisting tissue morphology.

There is a new developed a post-extraction fresh socket classification system as follows: Type 1: The facial soft tissue and buccal plate of bone are at normal levels in relation to the cement enamel junction of the pre-extracted tooth and remain intact post extraction.

Type 2: Facial soft tissue is present, but the buccal plate is partially missing following extraction of the tooth. Type 3: The facial soft tissue and the buccal plate of the bone are both markedly reduced after tooth extraction. This classification enabled ordering and classifying of post-extraction sockets.

A recently published sub-classification of type 2, now allows even greater clarity to plan regeneration: Type 2 A: Absence of the coronal one-third of labial bone plate of the extraction socket 5mm to 6mm from the free gingival margin. Type 2 B: Absence of the middle to coronal two thirds of the labial bone plate of the extraction socket approximately 7mm to 9mm from the free gingival margin.

Type 2 C: Absence of the apical one-third of the labial bone plate of the extraction socket 10 mm or more from the free gingival margin. For the management of socket defects after extraction numerous techniques have been developed to allow for optimum esthetic and functional outcomes. Among those techniques are ice cream cone technique described by Deniss Tarnow and the more recently introduce vestibular socket therapy (VST) introduced by Abd Salam Elaskary . Deniss Tarnow invented his technique (ice cream cone) to augment the socket with buccal dehiscence, in this technique, socket preservation was done using a collagen membrane shaped into an ice cream cone and placing it inside the extraction socket to cover the dehiscence site and the socket occlusally at the same time.

The regeneration of the buccal plate using the "ice cream cone" technique was possible in the dental extraction and by the immediate implant in an infected site in a case report of a 53 years old patient, and also in a clinical case series. But this technique is only recommended for simple dehiscence and not a wall defect. This technique is not applicable for a completely defective or missing bone wall unless a flap is raised, and (GBR) procedure is performed. Difficulty in placing the membrane as it become softened when exposed to fluid. In 2020 , Abd salam Elaskary , introduced vestibular socket therapy (VST), a novel minimally invasive surgical technique that allowed placement of immediate implant in maxillary class I and class II fresh extraction sockets with or without infective signs.

A 1-cm long vestibular access incision was made using a 15 blade 5-6 mm apical to the mucogingival junction of the socket, exposing the alveolar bone. The vestibular tissues were dissected in a coronal direction to detach the periosteum, forming a sub-periosteal tunnel connecting the vestibular incision to the socket orifice,bone graft was then introduced through the vestibular access incision to augment the labial plate of bone and fill any jumping gap. A flexible cortical membrane of 0.6 mm thickness was inserted and positioned 1 mm apical to the soft tissue margin and secured using two tacks apically. A customized healing abutment was fabricated to cover the implant and seal the socket .

This technique has many advantages : firstly, the nature of the vestibular extraction approach does not cause any trauma, pressure, or laceration to the soft tissue margin, which in turn has a positive impact on enhancing the mid-facial soft tissue levels, as the root was only pushed in an incisal direction through the created 6vestibular pouch, thus minimizing the osteoclastic activity around the socket rim .

, so it overcomes the remodeling sequelae of tooth extraction and to minimize the mid facial peri-implant gingival recession.

Secondly ,the use of a slowly resorbing flexible labial shield allowed for remodeling of the underlying labial bone plate while maintaining the socket dimensions and contours throughout the follow-up period. Thirdly, the membrane fixation, which is known to be pivotal for the GBR stability and regenerative outcomes. and finally connective tissue grafting can be done in type II sockets exhibiting a thin biotype. In these cases, the soft tissue graft counteracted the detrimental effect of the thin gingival phenotype on horizontal bone loss and midfacial mucosal recession.

VST can manage both type I and II socket defects, and could shorten the treatment time by up to two-thirds of that required for bone grafting and delayed implant placement.

ELIGIBILITY:
inclusion criteria :

1. Age more than 18 - 40 years.
2. Patients with missing single tooth or teeth in the esthetic zone.
3. Patients with buccal wall defect Type 2 A, B sockets (thin labial plate of bone less than 0.5 mm, presence of dehiscence or fenestration).
4. Good oral hygiene.
5. Patients willing to be present during the study follow-up intervals.
6. Patients free from any systemic diseases that may contraindicate implant placement .
7. Crown height space of at least 8 mm.
8. Patients without any para-functional habits (bruxism and clenching).

Exclusion Criteria:

1. Smoking people.
2. Alcohol or drug abuse.
3. Pregnancy.
4. Patients with poor oral hygiene or progressive periodontal disease .

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-04-21 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Bone changes | 12 months
  bone changes in volume by cone-beam computed tomography (CBCT )radiographically .

SECONDARY OUTCOMES:
soft tissue changes | 12 months
  evaluation of Probing depth around implants by a graduated dental probe , differences in volume changes by Standard Triangle Language( STL) files superimposition of the arches digitally by etc: Medit software.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarnachiaro GO, Chu SJ, Sarnachiaro E, Gotta SL, Tarnow DP. Immediate Implant Placement into Extraction Sockets with Labial Plate Dehiscence Defects: A Clinical Case Series. Clin Implant Dent Relat Res. 2016 Aug;18(4):821-9. doi: 10.1111/cid.12347. Epub 2015 Apr 27. PMID 25916859
- [Background] undefined
- [Background] Th Elaskary A, Gaweesh YY, El Tantawi M, Maebed MA. Vestibular Socket Therapy: A Novel Approach for Implant Placement in Defective Fresh Extraction Sockets With or Without Active Socket Infection (One-Arm Cohort Study). Int J Oral Maxillofac Implants. 2021 Jan-Feb;36(1):146-153. doi: 10.11607/jomi.8732. PMID 33600536
- [Background] Ghallab NA, Elaskary A, Elsabagh H, Toukhy AE, Abdelrahman H, El-Kimary G. A novel atraumatic extraction technique using vestibular socket therapy for immediate implant placement: a randomized controlled clinical trial. Oral Maxillofac Surg. 2023 Sep;27(3):497-505. doi: 10.1007/s10006-022-01089-4. Epub 2022 Jun 20. PMID 35718834
- [Background] Elaskary A, Meabed M, Abd-ElWahab Radi I. Vestibular socket therapy with immediate implant placement for managing compromised fresh extraction sockets: A prospective single-arm clinical study. Int J Oral Implantol (Berl). 2021 Aug 20;14(3):307-320. PMID 34415130
- See also: An Ice cream cone technique. Paper — https://pubmed.ncbi.nlm.nih.gov/26247445/